CLINICAL TRIAL: NCT03679299
Title: Vascular Implications of a Naturally Occurring Asthma Exacerbation
Status: Terminated | Type: Observational
Why Stopped: Poor study recruitment
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00083372
Record Dates: First submitted 2018-09-14; First posted 2018-09-20 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Asthma; Inflammation; Cardiovascular Risk Factor
Keywords: Flow-mediated dilation (FMD); arterial stiffness; pulse wave velocity (PWV); cardiovascular risk and asthma; endothelial function; systemic inflammation; C-reactive protein (CRP); eosinophils; neutrophils; asthma exacerbation
MeSH Terms: conditions — Asthma; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples collected for analysis of serum: systemic inflammation markers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Control: Healthy controls will be recruited from the general population and will be matched based on age, sex, and BMI. They will be assess at two time points, 48 hours apart. At each testing day, a blood sample will be taken, and endothelial function will be assessed using brachial artery flow mediated dilation. Arterial stiffness will be assessed using carotid-radial pulse wave velocity.
  Interventions: Other: Observational - No intervention
- Asthma: Individuals experiencing an asthma exacerbation will be recruited from the University of Alberta Hospital Emergency Department. Once discharged, a blood sample will be taken, and endothelial function will be assessed using brachial artery flow mediated dilation. Arterial stiffness will be assessed using carotid-radial pulse wave velocity. Participants will complete the same assessments at a follow up date 48 hours and 14 days post-discharge, with the addition of a full pulmonary function test, physical activity assessment via a Fitbit, and the completion of two questionnaires: Asthma Control Questionnaire, and Asthma Quality of Life Questionnaire.
  Interventions: Other: Observational - No intervention

INTERVENTIONS:
Other: Observational - No intervention — See outcomes

SUMMARY:
Although asthma is a disease of the airways, research is now showing that asthmatics are more likely to develop cardiovascular disease (CVD) compared to non-asthmatics. Vascular dysfunction is seen in people at high risk of CVD and has been linked to inflammation. During an asthma attack, levels of inflammation in the whole body increase, which could potentially explain why asthmatics are at increased risk of CVD. In the proposed study the investigators will examine if asthma attacks lead to increased risk of CVD by evaluating inflammatory levels and vascular function directly following asthma attacks, 2 days and 14 days after discharge. The investigators will compare these results to non-asthmatics. The results from this study will help us understand why asthmatics are at increased risk of CVD.

DETAILED DESCRIPTION:
BACKGROUND & SCOPE: While asthma is generally considered to be a disease of the airways, there are important systemic consequences which have predisposed people with asthma to become more likely to die from cardiovascular (CV) disease compared to non-asthmatics. Additional CV risks have been reported in people with severe asthma, and there is a relationship between reductions in lung function and cardiac death. To date, little is known in regards to the interaction between an asthma exacerbation and CV risk.

Brachial flow-mediated dilation (FMD) is used as a non-invasive tool to evaluate endothelial function. Brachial FMD is impaired in people with coronary dysfunction, and has been shown to predict future CV events better than traditional CV risk factors. People with asthma have previously been shown to have impaired endothelial function compared to non-asthmatics, but the underlying mechanism(s) are unclear. The aim of this study is to evaluate the endothelial function in people with asthma directly following an asthma exacerbation, 2 days and 14 days post-exacerbation, as well as non asthmatic controls.

Applanation tonometry is a non-invasive tool to evaluate arterial stiffness. It measure the pulse wave velocity (PWV), which is an independent predictor of cardiovascular risk. People with asthma have previously been shown to have increased arterial stiffness compared to non-asthmatics, but hte underlying mechanism(s) are unclear. Arterial stiffness will be evaluated in people with asthma directly following an asthma exacerbation, 2 days and 14 days post-exacerbation, as well as non asthmatic controls. Arterial stiffness, together with endothelial function will give information on the vascular function of the individuals.

Chronic systemic inflammation is an established risk factor and predictor of future CV events, and levels of systemic inflammation has been shown to be increased in asthma and to be are related to disease severity. While systemic inflammation can directly impair vascular function, it is unknown how an asthma attack may affect vascular function and CV risk. Thus, to gain better understanding of the increased CV risks associated with an asthma exacerbation, this study will evaluate the level of systemic inflammation in people with asthma directly following an asthma exacerbation, 2 days and 14 days post-exacerbation, as well as non asthmatic controls.

OBJECTIVE 1: To examine the vascular function and systemic inflammation in young adults experiencing a naturally occurring asthma exacerbation and to compare these data to values obtained from two follow up visits, as well as to healthy controls.

METHODS & PROCEDURES: Outline:

Each participant from the exacerbation group will be tested at three different times: Day 1) ED visit, Day 2) 48 hours post ED, Day 3) 14 days post ED.

A waist circumference measurement will be taken. Waist circumference will be measured at the level of the last rib to the nearest 0.1 cm after a normal expiration.

On Day 1, participants will be recruited by the Emergency Medicine Research Group (EMeRG). They will receive standard emergency care for their asthma and once stabilized, informed consent will be obtained. Once stabilized, the participant will be taken to a private area within the ED department to ensure no interference with ED procedures. Applanation tonometry will be done to measure PWV, followed by brachial FMD to determine endothelial function and lastly a blood sample will be obtained to measure serum CRP.

On Day 2 the participant will return and the same assessments as Day 1 will be performed with the addition of spirometry. A FitBit will be given along with instructions to wear the device for 7 days.

Day 3 will consist of the same measurements done in the ED for Day 1, with the addition of 2 quality of life questionnaires, the standardized Asthma Quality of Life Questionnaire (AQLQs) and the EQ-5D (5L), and the Asthma Control Questionnaire (ACQ), finishing with a pulmonary function test. Healthy controls will be tested two times, 48 hours apart. The same assessments as the exacerbation group will be done, but no FitBit or questionnaires will be given.

Spirometry: the participant will be tested for significant airway reversibility as per established clinical guidelines

Pulmonary function: A standard pulmonary function test will be performed by all participants as per established clinical guidelines.

Systemic inflammation and immune response markers present in venous blood samples will be analyzed at the University of Alberta.

Vascular function: Flow-mediated dilation (FMD) of the brachial artery following 5 minutes of forearm occlusion will be measured ultrasound imaging using our ultrasound machine. FMD will be determined using Doppler ultrasound immediately after the release of the occlusion. The secondary outcome is arterial stiffness, which will be determined using carotid - radial pulse wave velocity, and PWV will be calculated from measurements of pulse transit time and the distance traveled by the pulse between recording sites.

Physical Activity: will be measure with a FitBit activity monitored and calculated as average steps/day.

Questionnaires: will asses asthma control, disease specific quality of life, and generalized quality of life.

Data Analysis

The mean differences in FMD, systemic inflammation, and arterial stiffness for ED visit compared to the control group will be evaluated using an unpaired t-test. A within-factors repeated measures analysis of variance (ANOVA) will evaluate the mean differences between each assessment day for the exacerbation group to assess change in endothelial function during exacerbation as well as the recovery period. A similar evaluation will be used for arterial stiffness and systemic inflammation. A one-way analysis of covariance (ANCOVA) will be used to correct for shear rate in FMD for all groups, with both values being reported. A Pearson correlation will be used to determine any relationship between recovery rate and physical activity levels. In an exploratory sub analysis, unpaired t-tests will be used to evaluate the sex differences for each outcome.

An α-level of 0.05 will be used as the significance level for all statistical analysis, and all results will be reported as mean ± standard deviation unless indicated otherwise.While the impact of asthma exacerbations on vascular function is currently unknown, sample size calculations based on preliminary velocity-time integral (VTI) data from 11 confirmed asthmatics who underwent mannitol and placebo challenges indicate a total of 36 asthmatics and 36 controls would be sufficient to detect a 13% difference between these groups in VTI. Our preliminary data show a large increase in CRP in asthmatics experiencing an exacerbation vs. stable patients (7.3 vs. 0.5 mg/L, p<0.05), which would correspond to a substantial increase in CV risk, and be detectable with this sample size. An additional 8 participants per group will be recruited (i.e. 44 asthmatics and 44 controls) to compensate for potential dropouts. Sub-analyses evaluating potential sex-based differences will be exploratory and results will be considered hypothesis-generating.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18 and 55 years old
* waist circumference less than 88 cm for women and 102 cm for men.
* Asthma participants will be recruited from the University of Alberta Emergency Department with asthma exacerbation as their primary reason for visit.
* healthy controls will be recruited from the general population according to the same criteria, but with no history of asthma.

Exclusion Criteria:

* known heart failure or unstable cardiac disease,
* lung diseases other than asthma,
* known chronic inflammatory condition other than asthma
* known metabolic disease
* current infections,
* smoking history > 10 pack years,
* or waist circumference >88 cm for women and >102 cm for men

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Asthma participants recruited from the emergency department when seeking emergency care for an asthma exacerbation is the primary reason for visit.
  Healthy controls recruited from the general population.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Flow-mediated dilation | Emergency Department (ED), 48 hours and 14 days post ED for asthmatics, 2 time points 48 hours apart for controls.
  Percent change in diameter in response to shear stress

SECONDARY OUTCOMES:
C-reactive protein | Emergency Department (ED), 48 hours and 14 days post ED for asthmatics, 2 time points 48 hours apart for controls
  A marker for systemic inflammation and immune response
Eosinophils | Emergency Department (ED), 48 hours and 14 days post ED for asthmatics, 2 time points 48 hours apart for controls
  A marker for systemic inflammation and immune response
Neutrophils | Emergency Department (ED), 48 hours and 14 days post ED for asthmatics, 2 time points 48 hours apart for controls
  A marker for systemic inflammation and immune response
Pulse wave velocity | Emergency Department (ED), 48 hours and 14 days post ED for asthmatics, 2 time points 48 hours apart for controls
  Carotid radial arterial stiffness

OTHER OUTCOMES:
Average step count | Fitbit worn in asthmatics for 7 days following 48 hour timepoint
  Physical activity measured during first 2 weeks of recovery following an asthma exacerbation

CONTACTS AND LOCATIONS:
Overall Officials: Michael K Stickland, PhD, Principal Investigator — Professor, Division of Pulmonary Medicine, Department of Medicine; Director, G.F. MacDonald Centre for Lung Health Covenant Health; Scientific Director, Respiratory Health Strategic Clinical Network, Alberta Health Services
Locations (2):
- Canada (2):
  - University of Alberta Hospital Emergency Department, Edmonton, Alberta
  - Desi Fuhr, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/99/NCT03679299/Prot_SAP_001.pdf